CLINICAL TRIAL: NCT00265070
Title: An Open-Label, Phase II Trial Of 250 mg ZD1839 (IRESSA™) In Prostate Cancer Patients With Early Biochemical Failure Post Prostatectomy
Brief Title: Trial of Iressa in Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0093
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250 mg tablet oral daily dose
  Other Names: Iressa®; ZD1839

SUMMARY:
This study is being carried out to see if ZD1839 is effective in treating prostate cancer after being diagnosed with an early rising PSA (prostate specific antigen) following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Removal of prostate for prostate cancer
* Raised level of prostate specific antigen (PSA) post-surgery
* Can have received some radiation therapy

Exclusion Criteria:

* Any after surgery male hormone blocking therapy.
* Low white blood cell count
* Abnormal liver function test

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-01; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of the trial is to evaluate the activity of oral ZD1839 (250 mg once daily administered continuously) in subjects with early biochemical failure post prostatectomy by estimating the PSA response rate

SECONDARY OUTCOMES:
To estimate the duration of PSA response
To estimate the partial PSA response rate
To estimate the change in the ratio of free PSA : total PSA at 6 and 12 months compared with baseline
To investigate the change in PSA levels after discontinuation of ZD1839

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Canada Oncology Medical Director, MD, Study Director — AstraZeneca
Locations (4):
- Canada (4):
  - Research Site, Vancouver, British Columbia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal